CLINICAL TRIAL: NCT02298595
Title: A Phase I/II Study of BYL719, Cetuximab, and Cisplatin in Transorally Resectable, HPV-Associated Oropharyngeal Squamous Cell Carcinoma
Brief Title: Cetuximab, Cisplatin and BYL719 for HPV-Associated Oropharyngeal Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Julie E. Bauman, MD, MPH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Julie E. Bauman, MD, MPH, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-057; CBYL719XUS08T (Other: Novartis)
Record Dates: First submitted 2014-11-11; First posted 2014-11-24 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Squamous; Squamous Cell Carcinoma; Oropharyngeal Neoplasms; Oropharyngeal Cancer
Keywords: Carcinoma; Squamous; Oropharyngeal; HPV; Resectable
MeSH Terms: conditions — Carcinoma, Squamous Cell; Oropharyngeal Neoplasms; Carcinoma | interventions — Cisplatin; Cetuximab; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Low risk (Experimental): 3 cycles (3 weeks) of induction chemotherapy (cisplatin+paclitaxel+BYL719) followed by transoral resection (TORS or TLM) and then observation.
  Interventions: Drug: cisplatin; Drug: Cetuximab; Drug: BYL719
- 2: Intermediate risk (Experimental): 3 cycles (3 weeks) of induction chemotherapy (cisplatin+paclitaxel+BYL719) followed by transoral resection (TORS or TLM) and then Intensity Modulated Radiation Therapy (IMRT).
  Interventions: Drug: cisplatin; Drug: Cetuximab; Drug: BYL719
- 3: High risk (Experimental): 3 cycles (3 weeks) of induction chemotherapy (cisplatin+paclitaxel+BYL719) followed by transoral resection (TORS or TLM) and then Intensity Modulated Radiation Therapy (IMRT) + cisplatin.
  Interventions: Drug: cisplatin; Drug: Cetuximab; Drug: BYL719

INTERVENTIONS:
Drug: cisplatin — 75 mg/m2 IV day 1 of each cycle
  Other Names: Platinol; Cisplatinum
Drug: Cetuximab — XXXX day 1, 8, and 15 of each cycle
Drug: BYL719 — 200, 250, 300, or 350 mg/day by mouth every day

SUMMARY:
This study evaluates the combination of BYL719, cisplatin and cetuximab as induction chemotherapy prior to minimally-invasive transoral surgery (TORS or TLM) and selective lymph node dissection (SLND), followed by risk-adapted intensity-modulated radiation therapy (IMRT) in patients with transorally resectable, Stage III-IVa, HPV-associated oropharyngeal squamous cell carcinoma (OPSCC).

DETAILED DESCRIPTION:
HPV status and tobacco use are the major independent prognostic factors for patients with OPSCC. Patients with HPV-associated OPSCC have a favorable prognosis when treated with chemotherapy, radiation, and/or surgery. This has resulted in national trials investigating de-intensification strategies for good-risk patients with HPV-associated OPSCC, where current multimodality paradigms may represent overtreatment.

The PI3K/Akt/mTOR signaling network, a mitogenic pathway regulating cellular metabolism, proliferation and survival, plays a major role in HPV biology. Starting with early infection, activation of PI3K suppresses autophagy and induces functional protein translational machinery. Activation of the pathway is a nearly universal aspect of mammalian viral infection, and is of particular importance for dsDNA viruses such as HPV. The oncoproteins E5, E6 and E7 also have direct roles in pathway activation. Moreover, HPV-associated OPSCC demonstrates a strikingly high prevalence of genomic activation of the PI3K pathway, including activating PIK3CA mutations (27-31%), PIK3CA amplification (20%), and loss of PTEN (30%), the negative regulator of PI3K. Overall genomic events hypothesized to result in PI3K pathway activation are present in approximately 45-60% of HPV-transformed OPSCC.

BYL719 is an oral, small molecule, alpha-specific inhibitor of PI3-Kinase. Because HPV-associated OPSCC demonstrates a high rate of both genomic and non-genomic PI3K pathway activation, we hypothesize that adding BYL719 to platinum-taxane induction chemotherapy in HPV-associated OPSCC will increase clinico-radiologic complete response relative to historical control. In this phase I/II trial, eligible patients wiht HPV-associated OPSCC will be treated with 3 cycles of induction BYL719, cisplatin and paclitaxel. Induction will be followed by minimally-invasive, transoral surgery (TORS or TLM) then risk-adapted IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, cytologically or histologically confirmed squamous cell carcinoma (and common variants, including poorly differentiated carcinoma; undifferentiated carcinoma; basaloid carcinoma) of the oropharynx. Patients must have resectable oropharyngeal and nodal disease, including the following stages according to the American Joint Commission on Cancer Staging 7th edition:

  * T1N1-3
  * T2N1-3
  * T3N0-3
  * T4aN0-3. Note: Eligible T4a tumors may include deep/extrinsic tongue muscle invasion and must be judged resectable by TLM or TORS, according to the surgeon-investigator. Patients with T4a tumors with clear radiologic mandibular, hard palate or medial pterygoid invasion are not eligible.
* Carcinoma must be HPV-associated, which is defined as positive for p16 protein by immunohistochemistry (IHC). p16 positivity is defined as ≥70% of tumor cells demonstrating diffuse cytoplasmic and nuclear staining for p16 by immunohistochemistry in a CLIA certified pathology lab. p16 testing is standard at participating institutions and may be conducted locally.
* No evidence of distant metastatic disease
* Patients must have a clinically measurable primary oropharyngeal tumor, defined as measuring ≥ 1 cm by spiral CT, per RECIST 1.1, and/or by clinical examination.
* No prior systemic chemotherapy, systemic biologic/molecular targeted therapy or radiation treatment for head and neck cancer.
* Patients may have received chemotherapy or radiation for a previous, curatively treated non-HNSCC malignancy, provided at least 2 years have elapsed without evidence of recurrence.
* Patients must be untreated with radiation above the clavicles.
* Patients with a history of curatively-treated non-HNSCC malignancy must be disease-free for at least 2 years except for excised and cured: carcinoma-in-situ of breast or cervix; non-melanomatous skin cancer; T1-2, N0, M0 resected differentiated thyroid carcinoma; superficial bladder cancer; T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection.
* Age ≥ 18 years
* Patient has signed the Informed Consent Form (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements
* Patient has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1 that the investigator believes is stable at the time of screening
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤ 1.5
  * Creatinine Clearance ≥ 60 mg/mL as calculated by the modified Cockraft-Gault formula:

Calculated Creatinine Clearance = [(140-age) X (actual body weight in kg) X (0.85 if female)]/(72 X serum creatinine)

* Total serum bilirubin ≤ 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Fasting plasma glucose (FPG) ≤ 140mg/dL or ≤ 7.8 mmol/L

  * Patient is able to swallow and retain oral medication

Exclusion Criteria:

* Patient with poorly controlled diabetes mellitus, defined as FPG > 140 mg/dL or 7.8 mmol/L
* Patient has a history of another malignancy within 2 years prior to starting study treatment, except for excised and cured: carcinoma-in-situ of breast or cervix; non-melanomatous skin cancer; T1-2, N0, M0 differentiated thyroid carcinoma; superficial bladder cancer; T1a or T1b prostate cancer comprising < 5% of resected tissue with normal PSA since resection.
* The presence of distant metastatic disease
* Prior systemic chemotherapy, molecularly targeted therapy, or radiation therapy for the current OPSCC diagnosis
* History of radiation to the head and neck (above the clavicles)
* Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from side effects of such procedure.
* Patient has clinically significant cardiac disease or impaired cardiac function, such as:

  * Congestive heart failure (CHF) requiring treatment (New York Heart Association (NYHA) Grade ≥ 2), left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high-grade/complete AV-blockage
  * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), < 3 months prior to screening
* QT interval adjusted according to Fredericia (QTcF) > 480 msec on screening ECG
* Patient who has any severe and/or uncontrolled medical conditions such as:

  * Active or uncontrolled severe infection requiring systemic antibiotics or antifungals
  * Liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA)
  * Known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
  * Active bleeding diathesis
* Chronic treatment with corticosteroids or other immunosuppressive agents
* Chronic treatment with warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Grade ≥ 2 peripheral neuropathy
* Grade ≥ 2 sensorineural hearing loss
* Patient who is currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment.
* Patient who is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzymes CYP34A or CYP2C8. The patient must have discontinued moderate and strong inducers of either enzyme for at least one week and must have discontinued strong and moderate inhibitors before the start of treatment. Switching to a different medication prior to start of treatment is allowed.
* Patient with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, malabsorption syndrome, or small bowel resection).
* Patient with known positive serology for human immunodeficiency virus (HIV).
* Pregnant or nursing woman, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

  * Sexually active males should use a condom during intercourse while taking drug and for 12 weeks after completion of all protocol treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid, during the period of BYL719 treatment (induction chemotherapy) and for 4 weeks following completion of BYL719.
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and 12 weeks after completion of all study treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male partner sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of the following methods:
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Note: hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as BYL719 may decrease the effectiveness of hormonal contraceptives
  * Note: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Complete clinico-radiologic response of primary tumor following induction therapy | 10-11 weeks

SECONDARY OUTCOMES:
Pathologic response of primary tumor and lymph nodes following induction therapy | 16-19 weeks
2 year recurrence-free survival | 2 years
Duration of survival | 5 years
Proportion of patients with genomic PI3K pathway activation who have a complete clinico-radiologic and/or pathologic response to induction therapy | 10-13 weeks
  Genomic activation defined as: PIK3CA mutation, PIK3CA amplification, and/or PTEN deletion in baseline tumor
Number of participants with adverse events | 10-13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, MD, MPH, Principal Investigator — University of Pittsburgh